CLINICAL TRIAL: NCT05893563
Title: 5 Year Migration of Collared or Collarless Corail Stems Following THA
Brief Title: Corail Stability at 5-Years Post-Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Brent Lanting, Orthopaedic Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 13405
Record Dates: First submitted 2023-05-21; First posted 2023-06-08 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Total Hip Arthroplasty
Keywords: Implant Migration; Radiostereometric Analysis; CT Imaging; Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — microbial DNA in stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Direct Anterior: Patients who underwent the Direct Anterior (DA) surgical approach
  Interventions: Other: Standard Post-Operative Clinic Visit; Other: Study-Specific Outcomes
- Direct Lateral: Patients who underwent the Direct Lateral (DL) surgical approach
  Interventions: Other: Standard Post-Operative Clinic Visit; Other: Study-Specific Outcomes

INTERVENTIONS:
Other: Standard Post-Operative Clinic Visit — In clinic, the joint will be assessed (ROM, stability testing), standard X-rays will be taken of the joint, and patient reported outcomes (questionnaires) will be completed by patient (WOMAC, UCLA, VR12, EQ5D, Oxford Hip).
Other: Study-Specific Outcomes — Patients will complete additional questionnaires (SF12 and HHS), will undergo RSA and CT imaging for implant stability analysis, and will provide a stool sample for gut microbiome analysis.

SUMMARY:
Total hip arthroplasty (THA) is the mainstay, definitive management for end-stage hip osteoarthritis. Despite improvements of surgical and patient factors, prosthesis-related complications continue to increase in number. This is contributed to by the greater number of such surgeries being completed, larger proportion of elderly individuals among the population, and younger patient age being offered surgical intervention. Specifically, implant loosening and associated migration, is the pathology most commonly yielding revision surgery. A previous study assessing migration of total hip prostheses found that the greatest degree of migration occurred in the first 2 weeks postoperatively, although implants were considered overall stable 2 year following surgery. Continued evaluation of implant migration at time points further from surgery, specifically at 5 years postoperatively, offers insight into long term complications rates. Assessing implant migration will be completed using various imaging modalities, radiostereometric analysis (RSA) and computed tomography (CT). Comparisons between RSA and CT imaging will allow for greater analysis with regards to characterization of implant migration and associated bony changes. Additionally, an individual's gut microbiome has been shown to correspond to their inflammatory and immune profile. Association between gut microbiome profile and implant migration will be assessed to determine if underlying relationship does exist.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the originally investigated cohort.
* Minimum of 4-5 years post-operation

Exclusion Criteria:

* Pregnancy
* Unable to attend follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients previously recruited to a prospective RCT (NCT03558217), will be eligible to participate in this study. These patients were recruited preoperatively and underwent total hip arthroplasty using either the direct anterior or the direct lateral surgical approach. Each patient was also randomized to either receive a collared or collarless stem design. In the original study, patients were followed up until two-years postoperation, where the primary outcome measure was implant migration compared between surgical approach and implant design.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Implant Migration | at 5-years post-THA
  Measure implant migration that has occurred up until 5-years post-operation using RSA.

SECONDARY OUTCOMES:
WOMAC Score | at 5-years post-THA
  Assess the WOMAC clinical outcome questionnaire of the originally investigated cohort at 5 years post-operation compared to pre-surgery and early post-surgery.
SF12 Score | at 5-years post-THA
  Assess the SF-12 clinical outcome questionnaire of the originally investigated cohort at 5 years post-operation compared to pre-surgery and early post-surgery.
HSS Score | at 5-years post-THA
  Assess the HHS clinical outcome questionnaire of the originally investigated cohort at 5 years post-operation compared to pre-surgery and early post-surgery.
UCLA Score | at 5-years post-THA
  Assess the UCLA clinical outcome questionnaire of the originally investigated cohort at 5 years post-operation compared to pre-surgery and early post-surgery.
Inducible Displacement | at 5-years post-THA
  Compare the amount of inducible displacement measured between supine and weight bearing RSA and between internal and external rotation CT exams to validate the accuracy and precision of CT for implant migration analysis.
Joint Imaging Features | at 5-years post-THA
  Correlate CT-based measurements of bone density and texture features with the magnitude of implant migration using slicer (slicer.org) software to segment and analyze the CT images.
Gut Microbiome Analysis | at 5-years post-THA
  Correlate gut microbiome biomarkers for osteoporosis with the magnitude of implant migration by analyzing the microbial DNA in stool samples. The Shannon index for microbial diversity will be calculated and then correlated to the magnitude of migration.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Lanting, Principal Investigator — Lawson Health Science Centre
Locations (1):
- London Health Science Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No